CLINICAL TRIAL: NCT02098967
Title: A Multi-Center, Open-Label, First-in-Human, Phase I Dose-Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO6839921, An MDM2 Antagonist, Following Intravenous Administration in Patients With Advanced Malignancies, Including Acute Myeloid Leukemia (AML)
Brief Title: A Study of the Safety and Pharmacokinetics of RO6839921, An MDM2 Antagonist, in Patients With Advanced Cancers, Including Acute Myeloid Leukemia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP28903; RG7775 (Other: Roche)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Neoplasms, Myelogenous Leukemia, Acute
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid | interventions — RO6839921

ARMS (3):
- Acute myeloid leukemia patients (Experimental)
  Interventions: Drug: RO6839921
- Cohort 0 (Experimental)
  Interventions: Drug: RO6839921
- Solid tumor patients (Experimental)
  Interventions: Drug: RO6839921

INTERVENTIONS:
Drug: RO6839921 — Non-escalating IV doses given on Days 1-5 of Cycle 1.
  Arms: Cohort 0
Drug: RO6839921 — Escalating IV doses of RO6839921 in solid tumor patients. Dose escalation will be calculated using the new Continual Reassessment Method (nCRM). RO6839921 will be given on Days 1-5 of 28-day cycles. Treatment will continue until disease progression, unacceptable toxicity or study discontinuation.
  Arms: Solid tumor patients
Drug: RO6839921 — Escalating IV doses of RO6839921 in AML patients. Escalation will follow an adapted rolling 6 design. Starting dose </= dose inducing Grade 2 toxicity in patients with solid tumors. RO6839921 will be given on Days 1-5 of 28-day cycles. Treatment will continue until disease progression, unacceptable toxicity or study discontinuation.
  Arms: Acute myeloid leukemia patients

SUMMARY:
This open label, Phase I study of RO6839921 is a dose-escalation study with two arms. Prior to investigations in either arm, patients in a single cohort, Cohort 0, will receive non-escalating, intravenous (IV) doses of RO6839921 daily on Days 1-5 of a 28-day cycle. Interim PK and safety data from this cohort will be evaluated before initiating dose-escalation.

In arm A, RO6839921 will be given to patients with advanced solid tumor malignancies. In Arm B, RO6839921 will be given to patients with relapsed/refractory acute myeloid leukemia (AML). The arms will escalate independently. Escalation will begin in solid tumor patients (Arm A) in single patient cohorts, using a new Continual Reassessment Method (n-CRM). Escalation for AML patients will be initiated at or below the dose level that causes >/= Grade 2 hematologic side effects in Arm A. Escalation in AML patients will follow a rolling 6 design.

In both arms, RO6839921 will be administered by IV infusion on Days 1-5 of 28-day cycles.

There will be no intrapatient dose escalation. All patients may be treated until disease progression/relapse or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Cohort 0 and Arm A

* Patient must have histologically or cytologically confirmed advanced cancer for which standard cures or relieving measures either do not exist, are ineffective or are not acceptable to the patient.
* Measureable disease according to RECIST criteria version 1.1.
* ECOG performance status of 0 to 1.
* Adequate bone marrow function.

Arm B

* Patients with documented acute myeloid leukemia (AML), except for acute promyelocytic leukemia.
* Patients with relapsed/refractory AML or patients who have not received prior therapy who are high risk according to European LeukemiaNet (ELN) criteria.
* ECOG performance status of 0 to 2.

For Cohort 0, Arms A and B

* Life expectancy of >/= 12 weeks.
* Age >/= 18 years or older.
* All patients must be willing to use effective methods of contraception until 10 days after the last dose; women must not be pregnant or breast-feeding.
* Adequate renal and hepatic function.
* Patients with stable central nervous system (CNS) tumors are eligible.
* There are no requirements or limitations on the amount or type of prior anti-tumor/anti-leukemia therapy.

Exclusion Criteria:

Cohort 0 and Arm A

* Patients with a history of any form of leukemia except for Stage 0 and 1 chronic lymphocytic leukemia (CLL) not requiring treatment.
* Patients receiving any cancer treatment within 21 days of start of study medication. Patients must also have recovered from severe side effects due to prior treatment before study start.
* Patients with known bone marrow disorders that may interfere with bone marrow recovery, or patients with delayed recovery from prior chemoradiotherapy.
* Patients with known bleeding or clotting disorders or non-drug-induced low platelet count.

Arm B

- Patients receiving any cancer treatment within 14 days of start of study medication. Hydroxyurea may be taken until first administration of the study drug. Patients must also have recovered from severe side effects due to prior treatment before study start.

For Cohort 0, Arms A and B

* Patients receiving any other test drugs within 30 days of start of study medication
* Patients receiving the cytochrome P450 inhibitors, substrates or inducers specified in the protocol.
* Anticoagulation or antiplatelet treatment must be discontinued 7 days prior to start of study medication.
* Patients who have received hormonal therapy (except for prostate cancer treatment and hormone replacement therapy) within the 2 weeks prior to start of study medication.
* Patients with evidence of electrolyte imbalance, which may be treated to meet eligibility.
* Serum albumin < 2.8 g/dL.
* HIV-positive patients who are currently receiving combination antiretroviral therapy.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Approximately 1 year
Incidence of dose-limiting toxicities | Approximately 1 year

SECONDARY OUTCOMES:
Plasma area under the concentration-time curve (AUC) of RO6839921. | Up to Day 22
Changes in serum macrophage inhibitory cytokine-1 (MIC-1) expression measured by enzyme-linked immunosorbent assay (ELISA) | Up to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (3):
  - University of Colorado, Aurora, Colorado
  - Washington University, St Louis, Missouri
  - Medical University of South Carolina; Hollings Cancer Center, Charleston, South Carolina
- Canada (2):
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Jewish General Hospital / McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Uy GL, Assouline S, Young AM, Blotner S, Higgins B, Chen LC, Yee K. Phase 1 study of the MDM2 antagonist RO6839921 in patients with acute myeloid leukemia. Invest New Drugs. 2020 Oct;38(5):1430-1441. doi: 10.1007/s10637-020-00907-4. Epub 2020 Feb 4. PMID 32020437
- [Derived] Abdul Razak AR, Miller WH Jr, Uy GL, Blotner S, Young AM, Higgins B, Chen LC, Gore L. A phase 1 study of the MDM2 antagonist RO6839921, a pegylated prodrug of idasanutlin, in patients with advanced solid tumors. Invest New Drugs. 2020 Aug;38(4):1156-1165. doi: 10.1007/s10637-019-00869-2. Epub 2019 Nov 16. PMID 31734832